CLINICAL TRIAL: NCT00365677
Title: Compare the Safety and Effectiveness of Two Versions of the Bausch & Lomb Zyoptix™ Tissue Saving Aspheric Algorithm to the Current Zyoptix™ Tissue Saving Algorithm When Used for Myopia and Myopic Astigmatism Lasik Treatment
Brief Title: A Study to Investigate the Safety and Effectiveness of Aspheric Laser Refractive Surgery Treatments for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 441
Record Dates: First submitted 2006-06-30; First posted 2006-08-17 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zyoptix Tissue Saving Aspheric (Experimental): The Bausch & Lomb Zyoptix Tissue Saving Aspheric algorithm is used for treatment with LASIK for the correction of myopia and myopic astigmatism.
  Interventions: Device: The Bausch & Lomb Zyoptix Tissue Saving Aspheric algorithm
- Zyoptix Tissue Saving (Active Comparator): The Bausch & Lomb Zyoptix Tissue Saving algorithm is used for treatment with LASIK for the correction of myopia and myopic astigmatism.
  Interventions: Device: The Bausch & Lomb Zyoptix Tissue Saving algorithm

INTERVENTIONS:
Device: The Bausch & Lomb Zyoptix Tissue Saving Aspheric algorithm — Used with LASIK treatment for the correction of myopia and myopic astigmatism.
  Arms: Zyoptix Tissue Saving Aspheric
Device: The Bausch & Lomb Zyoptix Tissue Saving algorithm — Used with LASIK treatment for the correction of myopia and myopic astigmatism.
  Arms: Zyoptix Tissue Saving

SUMMARY:
The objective of this study was to compare the safety and effectiveness of two versions of the Bausch & Lomb Zyoptix Tissue Saving Aspheric Algorithm versus the current Zyoptix Tissue Saving Algorithm when used for myopia and myopic astigmatism LASIK treatment.

ELIGIBILITY:
Inclusion Criteria:

* Myopia with or without astigmatism.
* Normal Corneal topography
* Willing to have both eyes treated with the laser.

Exclusion Criteria:

* Contraindications to LASIK.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity | At 90 days post surgery
Preservation of best spectacle corrected high contrast logMAR distance visual acuity compared to baseline. | At 90 days post surgery

SECONDARY OUTCOMES:
Deviation from target correction | At 90 days post surgery
Improvement in uncorrected distance high contrast logMAR visual acuity compared to baseline | At 90 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Egamino, PhD, Study Director — Bausch & Lomb Incorporated